CLINICAL TRIAL: NCT02803879
Title: Assessing the Capability of Cardiogoniometry (CGM) to Detect Changes in Cardiac Resynchronisation Therapy Device Settings
Acronym: HF-CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/NW/0479
Record Dates: First submitted 2016-02-18; First posted 2016-06-17 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: cardiac resynchronisation therapy; cardiogoniometry
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiogoniometry (CGM) (Experimental): All patients attending clinic for follow up appointments following the implantation of a CRT device will be eligible for inclusion in the study. If they consent for enrolment in the study each patient will undergo a series of 4 CGM recordings whilst in their follow up appointment. They will undergo each of these during different pacemaker settings. These are: 1) No pacing, 2) Paced from the right ventricular lead; 3) Paced from the left ventricular lead and 4) Paced from both ventricular leads. After this has been done the participants involvement in the study will have finished.
  Interventions: Device: Cardiogoniometry

INTERVENTIONS:
Device: Cardiogoniometry

SUMMARY:
Some patients with heart failure require treatment called cardiac-resynchronisation therapy (CRT) which involves putting a pacemaker into the heart to make both ventricles (the lower chambers of the heart) contract together, making the pumping of the blood to the rest of the body more efficient.

it is important to get the CRT pacemaker checked to make sure that it is working correctly and performing its job. However, it can be difficult to adjust the settings of the pacemaker just the right amount to ensure the heart is pumping efficiently.

One of the ways this can be done is by using a special machine which uses ultrasound to make a 2-dimensional image of the heart called an echocardiogram. This technique can also be used to measure the flow of blood in the heart and calculate how efficient it is at pumping blood. However adjusting the settings of the pacemaker with this device is difficult to use and time consuming.

Electrocardiogram (ECG) a 2-dimensional electrical tracing of the hearts activity is another tool used to help adjust the settings of pacemakers, to make the heart pump more efficiently. Furthermore, recent research has shown that this is better than echocardiogram at optimising pacemaker device settings.

A new type of ECG called cardiogoniometry (CGM) has recently been developed which creates a 3-dimensional view of the hearts electrical activity and has already been shown to be better than normal ECG at diagnosing certain conditions like angina and heart attacks. However it has never been used to try optimise the settings of the pacemakers used in CRT and may be quicker and easier to use than then other methods available. More importantly it is hoped by doing this it will reduce the symptoms that patients suffer as it is making the heart pump more efficiently.

As it has been untested and never used in this setting before, and there it is necessary to find out if the CGM machine will recognise when the settings on the pacemaker are changed.

The aims of this study is to see if the CGM machine can pick up changes to pacemaker settings, with the hope of running a later study to see if it can be used to optimise settings on the pacemaker used in CRT.

DETAILED DESCRIPTION:
Cardiac resynchronisation therapy (CRT) improves symptoms and quality of life and improves the prognosis of patients with chronic heart failure. CRT works by improving co-ordination of cardiac contraction, and is indicated in people with heart failure and left bundle branch block (LBBB) on an ECG. The importance of LBBB is that it indicates that the electricity is spreading only very slowly over the surface of the heart with each heart beat, thereby making contraction very "dyssynchronous"; that is, instead of all the heart muscle contracting simultaneously, parts contract and are relaxing before other parts even start to contract.

With a standard pacemaker, a pacing lead is implanted in the right ventricle. In those patients with a normal heart rhythm ("sinus rhythm"), a second lead is usually placed in the right atrium close to the heart's natural pacemaker. The lead in the ventricle can then track the heart's natural heart rate as detected by the lead in the atrium, or, if the natural rate is too slow, the pacemaker can sequentially pace the atrium and then the ventricle.

A CRT system is similar, but with the addition of an extra lead positioned to pace the left ventricle. Now, the pacemaker is able to stimulate both left and right ventricles simultaneously, restoring the normal co-ordination of ventricular contraction.

Approximately 25% of patients do not achieve significant clinical benefit with CRT. Such patients are termed "non-responders", and lack of response is typically measured as a failure to improve exercise capacity with CRT, or a failure of the heart to improve on echocardiography. One option to reduce the number of non-responders may be to optimise the CRT device by adjusting its settings based on clinical variables (such as ECG and echocardiogram findings). Both ECG and echocardiogram optimisation give similar results in terms of clinical response to CRT, but patients who had their CRT optimised using ECG variables had a significantly greater impact on echocardiographic response, that is a greater proportion of that group had a LV end-systolic volume reduction >10%) 3. Another possibility for optimising CRT is cardiogoniometry (CGM), which is what the study aims to investigate. CGM is form of 3D vector electrocardiography which can provide quantitative analysis of myocardial depolarisation and repolarisation. Like standard 12 lead electrocardiogram (ECG), CGM uses different electrodes to identify electrical potential gradients produced by cardiac electrical activity. The ECG can only visually represent this information in a two dimensional way, whereas CGM can create a three dimensional display. Electrode placement is important: and complex mathematical modelling is used to generate the displays. CGM gives the same output as a standard ECG. One additional output is vector loop graphs. These are sequentially plotted values of electrical activity of the heart in the x, y and z axis, in three orthogonal planes. When the vector loops follow the same pathway it means that the electrical activity of the heart is following the same pathway with each ventricular depolarisation and repolarisation. By contrast, when there is abnormal electrical conduction, the vector loop pathways can vary. CGM is useful for identifying stable coronary artery disease and recognising the acute coronary syndromes, but its clinical value outside patients with acute ischaemic heart disease is unclear. This feasibility study aims to see if CGM can detect the different settings of a CRT device, by assessing the CGM vector loops with different device settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending follow up clinic with a CRT device implanted.
* Patients have to be receiving CRT therapy - in other words, the device has to be functioning correctly.
* Aged 18 or over.
* The patient has been informed of the nature of the study and has provided full written informed consent.

Exclusion Criteria:

* Patients unable to give informed consent including those with communication difficulties due to poor English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean cardiac axis with no pacing | Within the first 30 days after end of participant enrollment
  Mean cardiac axis of participants when they are not being paced will be calculated with 95% confidence intervals.
Mean cardiac axis with rv pacing | Within the first 30 days after end of participant enrollment
  Mean cardiac axis of participants when they are being paced from the RV will be calculated with 95% confidence intervals.
Mean cardiac axis with lv pacing | Within the first 30 days after end of participant enrollment
  Mean cardiac axis of participants when they are being paced from the LV will be calculated with 95% confidence intervals.
Mean cardiac axis with biv pacing | Within the first 30 days after end of participant enrollment
  Mean cardiac axis of participants when they are being biventricular paced will be calculated with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brown OI, Nikolaidou T, Beddoes G, Hoye A, Clark AL. The HF-CGM Study: An Analysis of Cardiogoniometric Axes in Patients With Cardiac Resynchronization Therapy. IEEE Trans Biomed Eng. 2018 Aug;65(8):1711-1716. doi: 10.1109/TBME.2017.2769060. Epub 2017 Nov 2. PMID 29989935
- See also: Abstract Link — https://www.ncbi.nlm.nih.gov/pubmed/29989935?dopt=Abstract